CLINICAL TRIAL: NCT02942836
Title: CareTaker Respiratory Rate Detection Study
Acronym: RSP
Status: Completed | Type: Observational
Sponsor: CareTaker Medical LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: RSP_001
Record Dates: First submitted 2016-10-20; First posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Respiration Rate Detection
Keywords: Respiration Rate Detection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: non-intrusive respiration monitor — Equivalence of CareTaker's respiration rate detection capability to that of predicate device

SUMMARY:
The goal of the proposed study is to test the capability of the CareTaker monitor to extract the respiration signature from its acquired signal, and to determine a respiration rate of breaths/minute that meets or exceeds the performance levels of its predicate device.

DETAILED DESCRIPTION:
The goal of the proposed study is to test the capability of the CareTaker monitor to extract the respiration signature from its acquired signal, and to determine a respiration rate of breaths/minute that meets or exceeds the performance levels of its predicate device.

The detection approach of RSPR (respiratory rate) that the CareTaker technology takes is based on peak detection and pulse analysis of arterial pressure pulse signals, as well as spectral analysis of the raw CareTaker sensor signal.

The study was performed under the supervision of the Chesapeake IRB and involved 21 subjects >18 y who were monitored during spontaneous and metronome-paced breathing.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age, who are able and willing to participate and have given verbal assent

Exclusion Criteria:

* Unable to give written consent
* <18 years of age
* No or poor finger pulse, as determined through visual inspection for ischemic hands

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects were local health club members, > 18 years of age, who were able and willing to participate and willing to sign the written consent
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Respiration rate detection with accuracy of better than 3 breaths per minute | 15 minutes of matched respiration rates
  Comparison with performance of predicate device (accuracy within 3 breaths per minute).

CONTACTS AND LOCATIONS:
Overall Officials: Martin C Baruch, PhD, Principal Investigator — CareTaker Medical LLC

IPD SHARING:
Plan to Share IPD: Undecided